CLINICAL TRIAL: NCT01774721
Title: ARCHER 1050: A RANDOMIZED, OPEN-LABEL, PHASE 3, EFFICACY AND SAFETY STUDY OF DACOMITINIB (PF-00299804) VERSUS GEFITINIB FOR THE FIRST LINE TREATMENT OF LOCALLY ADVANCED OR METASTATIC NON-SMALL CELL LUNG CANCER IN SUBJECTS WITH EPIDERMAL GROWTH FACTOR RECEPTOR (EGFR) ACTIVATING MUTATION(S)
Brief Title: ARCHER1050: A Study of Dacomitinib vs. Gefitinib in 1st-Line Treatment Of Advanced NSCLC.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: A7471050; DP312804 (Other: Pfizer)
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-01

CONDITIONS: Non-small Cell Lung Cancer With EGFR-Activating Mutations
Keywords: first-line; locally advanced or metastatic; non-small cell lung cancer; epidermal growth factor receptor; EGFR; ARCHER; mutation; dacomitinib; PF-00299804
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dacomitinib (PF-00299804) (Experimental): Dacomitinib (PF-00299804) is provided as 45 mg tablets, continuous oral daily dosing.
  Interventions: Drug: Dacomitinib (PF-00299804)
- gefitinib (Active Comparator): Gefitinib is provided as 250 mg tablets, continuous oral daily dosing.
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Dacomitinib (PF-00299804) — Dacomitinib (PF-00299804) 45 mg tablets, continuous oral daily dosing.
  Other Names: Dacomitinib
  Arms: Dacomitinib (PF-00299804)
Drug: Gefitinib — Gefitinib 250 mg tablets, continuous oral daily dosing.
  Other Names: Iressa
  Arms: gefitinib

SUMMARY:
This is a multinational, multicenter, randomized, open-label, Phase 3 study comparing the efficacy and safety of treatment with dacomitinib (PF-00299804) to treatment with gefitinib in patients with locally advanced or metastatic non-small cell lung cancer, with epidermal growth factor receptor EGFR-activating mutation (s). Analyses of primary objective (Progression Free Survival) will be done as defined in the protocol.

DETAILED DESCRIPTION:
452 patients were randomized in a 1:1 ratio between dacomitinib (PF-00299804 ) vs. gefitinib.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of histo or cytopathology confirmed, advanced NSCLC (with known histology) with the presence of EGFR-activating mutation (exon 19 deletion or the L858R mutation in exon 21).
* It is acceptable for subjects with the presence of the exon 20 T790M mutation together with either EGFR-activating mutation (exon 19 deletion or the L858R mutation in exon 21) to be included in this study
* No prior treatment with systemic therapy for locally advanced or metastatic NSCLC. Minimum of 12 months disease free interval between completion of neoadjuvant/adjuvant systemic therapy and recurrence of NSCLC
* Adequate tissue sample must be available for central analyses.
* Adequate renal, hematologic, liver function.
* ECOG PS of 0-1.
* Radiologically measurable disease.

Exclusion Criteria:

* Any evidence of mixed histology that includes elements of small cell or carcinoid lung cancer.
* Any other mutation other than exon 19 deletion or L858R in exon 21, with or without the presence of the exon 20 T790M mutation.
* Any history of brain metastases or leptomeningeal metastases.
* Any previous anti-cancer systemic treatment of early, locally advanced, or metastatic NSCLC.
* Any surgery(not including minor procedures such as lymph node biopsy), palliative radiotherapy or pleurodesis within 2 weeks of baseline assessments
* Any clinically significant gastrointestinal abnormalities that may impair intake, transit or absorption of the study drug.
* Current enrollment in another therapeutic clinical study.
* History of, or currently suspected, diffuse non-infectious pneumonitis or interstitial lung disease
* Uncontrolled medical disorders.
* Prior malignancy and concurrent malignancy except for non melanoma skin cancer or in-situ cervical cancer with no evidence of active disease.
* Use of narrow therapeutic index drugs that are CYP2D6 substrates from screening to randomization.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2013-05-09 (Actual); Primary Completion 2016-07-29 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- China (15):
  - Beijing
  - Changchun
  - Changsha
  - Chengdu
  - Chongqing
  - Fuzhou
  - Guangzhou
  - Hangzhou
  - Hefei
  - Nanning
  - Shanghai
  - Shenyang
  - Tianjin
  - Wuhan
  - Wuxi
- Hong Kong (2):
  - Hong Kong
  - Shatin
- Italy (11):
  - Catania
  - Lecco
  - Livorno
  - Meldola
  - Milan
  - Napoli
  - Perugia
  - Ravenna
  - Roma
  - Trento
  - Viterbo
- Japan (9):
  - Hokkaido, Asahikawa
  - Kashiwa, Chiba
  - Matsuyama, Ehime
  - Yokohama, Kanagawa
  - Tokyo, Koto-ku
  - Sakai, Osaka
  - Sayama, Osaka
  - Sunto-gun, Shizouka
  - Chuo-Ku, Tokyo
- Poland (4):
  - Gdansk
  - Olsztyn
  - Poznan
  - Warsaw
- Seoul, South Korea
- Spain (10):
  - Ávila
  - Barcelona
  - Bilbao
  - Cáceres
  - Córdoba
  - Donostia / San Sebastian
  - Las Palmas
  - Madrid
  - Málaga
  - Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Pu X, Li J, Zhang B, Zhang J, K Mok TS, Nakagawa K, Rosell R, Cheng Y, Zhou X, Miglorino MR, Niho S, Lee KH, Corral J, Pluzanski A, Li J, Linke R, Pan F, Tang Y, Tan W, Wu L. Efficacy in patients with EGFR-positive non-small-cell lung cancer treated with dacomitinib who had skin adverse events: post hoc analyses from ARCHER 1050. Future Oncol. 2024;20(37):2971-2982. doi: 10.1080/14796694.2024.2404762. Epub 2024 Oct 3. PMID 39360943
- [Derived] Li J, Nickens D, Wilner K, Tan W. Evaluation of the Effect of Proton Pump Inhibitors on the Efficacy of Dacomitinib and Gefitinib in Patients with Advanced Non-Small Cell Lung Cancer and EGFR-Activating Mutations. Oncol Ther. 2021 Dec;9(2):525-539. doi: 10.1007/s40487-021-00156-2. Epub 2021 Jun 13. PMID 34120312
- [Derived] Cheng Y, Mok TS, Zhou X, Lu S, Zhou Q, Zhou J, Du Y, Yu P, Liu X, Hu C, Lu Y, Zhang Y, Lee KH, Nakagawa K, Linke R, Wong CH, Tang Y, Zhu F, Wilner KD, Wu YL. Safety and efficacy of first-line dacomitinib in Asian patients with EGFR mutation-positive non-small cell lung cancer: Results from a randomized, open-label, phase 3 trial (ARCHER 1050). Lung Cancer. 2021 Apr;154:176-185. doi: 10.1016/j.lungcan.2021.02.025. Epub 2021 Feb 23. PMID 33721611
- [Derived] Mok TS, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Chawla A, Rosell R, Corral J, Migliorino MR, Pluzanski A, Noonan K, Tang Y, Pastel M, Wilner KD, Wu YL. Updated Overall Survival in a Randomized Study Comparing Dacomitinib with Gefitinib as First-Line Treatment in Patients with Advanced Non-Small-Cell Lung Cancer and EGFR-Activating Mutations. Drugs. 2021 Feb;81(2):257-266. doi: 10.1007/s40265-020-01441-6. PMID 33331989
- [Derived] Corral J, Mok TS, Nakagawa K, Rosell R, Lee KH, Migliorino MR, Pluzanski A, Linke R, Devgan G, Tan W, Quinn S, Wang T, Wu YL. Effects of dose modifications on the safety and efficacy of dacomitinib for EGFR mutation-positive non-small-cell lung cancer. Future Oncol. 2019 Aug;15(24):2795-2805. doi: 10.2217/fon-2019-0299. Epub 2019 Jul 17. PMID 31313942
- [Derived] Nagano T, Tachihara M, Nishimura Y. Dacomitinib, a second-generation irreversible epidermal growth factor receptor tyrosine kinase inhibitor (EGFR-TKI) to treat non-small cell lung cancer. Drugs Today (Barc). 2019 Apr;55(4):231-236. doi: 10.1358/dot.2019.55.4.2965337. PMID 31050691
- [Derived] Mok TS, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Lee M, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Wu YL. Improvement in Overall Survival in a Randomized Study That Compared Dacomitinib With Gefitinib in Patients With Advanced Non-Small-Cell Lung Cancer and EGFR-Activating Mutations. J Clin Oncol. 2018 Aug 1;36(22):2244-2250. doi: 10.1200/JCO.2018.78.7994. Epub 2018 Jun 4. PMID 29864379
- [Derived] Wu YL, Cheng Y, Zhou X, Lee KH, Nakagawa K, Niho S, Tsuji F, Linke R, Rosell R, Corral J, Migliorino MR, Pluzanski A, Sbar EI, Wang T, White JL, Nadanaciva S, Sandin R, Mok TS. Dacomitinib versus gefitinib as first-line treatment for patients with EGFR-mutation-positive non-small-cell lung cancer (ARCHER 1050): a randomised, open-label, phase 3 trial. Lancet Oncol. 2017 Nov;18(11):1454-1466. doi: 10.1016/S1470-2045(17)30608-3. Epub 2017 Sep 25. PMID 28958502
- [Derived] Ramalingam SS, O'Byrne K, Boyer M, Mok T, Janne PA, Zhang H, Liang J, Taylor I, Sbar EI, Paz-Ares L. Dacomitinib versus erlotinib in patients with EGFR-mutated advanced nonsmall-cell lung cancer (NSCLC): pooled subset analyses from two randomized trials. Ann Oncol. 2016 Mar;27(3):423-9. doi: 10.1093/annonc/mdv593. Epub 2016 Jan 13. PMID 26768165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study completed enrollment on 25 Mar 2015 with 452 participants randomized, 227 participants to the dacomitinib arm and 225 participants to the gefitinib arm. After the last data cutoff (DCO) date of 13 May 2019, 11 participants remained in the study to continue dacomitinib treatment. All 11 participants were discontinued from the study by last participant last visit (LPLV) on 27 Jan 2022.
Groups:
- Dacomitinib: Participants received 45 mg of dacomitinib tablets orally once daily in each treatment cycle of 28 days, up to a maximum of 48 months until disease progression, intolerable toxicities, withdrawal, death, or investigator decision dictated by protocol compliance, whichever occurred first.
- Gefitinib: Participants received 250 mg of gefitinib tablets orally once daily in each treatment cycle of 28 days, for maximum of 48 months until disease progression, intolerable toxicities, withdrawal, death, or investigator decision dictated by protocol compliance, whichever occurred first.
Period: Overall Study
Arm/Group | Dacomitinib | Gefitinib
Started | 227 | 225
Treated | 227 | 224
Completed | 0 | 0
Not Completed | 227 | 225
Not completed — Death | 133 | 152
Not completed — Withdrawal by Subject | 20 | 14
Not completed — Lost to Follow-up | 6 | 7
Not completed — Did not meet eligibility criteria | 0 | 3
Not completed — Other reasons and patients who completed the 48-month follow-up period | 58 | 49
Not completed — Study terminated by sponsor | 5 | 0
Not completed — Disease progression | 5 | 0

BASELINE CHARACTERISTICS:
Population: ITT Population included all participants who were randomized, with study treatment assignment designated according to initial randomization, regardless of whether participants received study treatment or received a different treatment from that to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dacomitinib | Gefitinib | Total
Number analyzed (Participants) | 227 | 225 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (11.26) | 60.9 (10.17) | 61.1 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 125 | 271
  Male | 81 | 100 | 181
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 227 | 225 | 452
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 170 | 176 | 346
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 56 | 49 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Independent Radiologic Central (IRC) Review
Description: PFS: time from randomization to date of progression of disease (PD) as determined by IRC review as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria or death due to any cause, whichever occurred first. PD: >=20% increase in sum of diameters of target lesions (TLs), referring smallest sum on study, sum must be an absolute increase of >=5 mm, appearance of >=1 new lesions; unequivocal progression of existing non TLs. Overall tumor burden increased sufficiently to merit discontinuation of therapy. In presence of stable disease (did not achieve partial response, complete response or PD) or partial response (>=30% decrease under baseline of sum of diameters of all target measurable lesions, short diameter used in the sum for target nodes, longest diameter used in sum for all other target lesions) in target disease; for new lesions: appearance of any new unequivocal malignant lesion indicated PD.
Time Frame: Day 28 of Cycle 1, Cycle 2 then every 8 weeks until disease progression or death due to any cause, whichever occurred first (up to 48 months)
Population: Intent to treat (ITT) Population included all randomized participants, with study treatment assignment designated according to initial randomization, regardless of whether participants received study treatment or a different treatment from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
months | 14.7 [11.1 to 16.6] | 9.2 [9.1 to 11.0]
Statistical Analysis 1: Comparison: Dacomitinib vs Gefitinib; Test type: Superiority; p < 0.0001, 1-sided stratified log-rank test; Hazard Ratio (HR) = 0.589, 95% CI 2-sided [0.469 to 0.739] — Based on stratified Cox regression model

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to the date of death for any cause. In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive. OS (month)=[death date or last known alive date - randomization date + 1]/30.4375.
Time Frame: From randomization until death or last date known as alive, up to 45 months
Population: ITT Population included all randomized participants, with study treatment assignment designated according to initial randomization, regardless of whether participants received study treatment or a different treatment from that to which they were randomized.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
months | 34.1 [29.5 to 39.8] | 27.0 [24.4 to 31.6]
Statistical Analysis 1: Comparison: Dacomitinib vs Gefitinib; Test type: Superiority; p = 0.0077, 1-sided stratified log-rank test; Hazard Ratio (HR) = 0.748, 95% CI 2-sided [0.591 to 0.947] — Based on stratified Cox Regression model

3. Secondary Outcome: OS at 30 Months (OS30m)
Description: OS30m was defined as the probability of a participant being alive at 30 months from date of randomization.
Time Frame: Up to 30 months from date of randomization
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
probability of survival | 56.4 [49.6 to 62.7] | 45.7 [39.0 to 52.2]

4. Secondary Outcome: Progression Free Survival (PFS) Based on Investigator Assessment
Description: PFS: time from randomization to date of PD as determined by investigator assessment as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria or death due to any cause, whichever occurred first. PD for target lesions: 20% increase in sum of diameters of target measurable lesions above smallest sum observed, with minimum absolute increase of 5 mm; for non-target lesions: unequivocal progression of pre-existing lesions. Overall tumor burden increased sufficiently to merit discontinuation of therapy. In presence of stable disease (did not achieve partial response, complete response or PD) or partial response (>=30% decrease under baseline of sum of diameters of all target measurable lesions, short diameter used in the sum for target nodes, longest diameter used in sum for all other target lesions) in target disease; for new lesions: appearance of any new unequivocal malignant lesion indicated PD.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gefitinib: Participants received 250 mg of gefitinib tablets orally once daily in each treatment cycle of 28 days, up to a maximum of 48 months until disease progression, intolerable toxicities, withdrawal, death, or investigator decision dictated by protocol compliance, whichever occurred first.
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
months | 16.6 [12.9 to 18.4] | 11.0 [9.4 to 12.1]
Statistical Analysis 1: Comparison: Dacomitinib vs Gefitinib; Test type: Superiority; p < 0.0001, 1-sided stratified log-rank test; Hazard Ratio (HR) = 0.622, 95% CI 2-sided [0.497 to 0.779] — Based on stratified Cox regression model

5. Secondary Outcome: Number of Participants With Best Overall Response (BOR) Based on IRC Review
Description: BOR for CR/PR:>=1 objective status (OBS) of CR/PR documented before PD; SD:>=1 OBS of stable documented >=8 weeks (wks) post treatment & before PD, not qualifying as CR/PR; PD:OBS of PD within 12 wks treatment, not qualifying as CR/PR/SD; indeterminate:PD not documented within 12 wks post treatment & no other response category applies. RECIST v1.1, CR:disappearance of all target lesions (TLs), non TLs;any pathological lymph nodes (LN) must reduce in short axis to <10 mm; normalization of tumour marker level, for non TL all LN must be non-pathological in size (<10 mm short axis); PR:>=30% decrease in sum of diameters of TLs, referring baseline sum diameters. SD:neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, referring smallest sum diameters on study. PD:>=20% increase in sum of diameters of TLs, referring smallest sum on study, sum must be an absolute increase of >=5 mm, appearance of >=1 new lesions;unequivocal progression of existing non TLs.
Time Frame: Day 28 of Cycle 1, Cycle 2 then every 8 weeks until disease progression (up to 48 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
Participants
  Complete response | 12 | 4
  Partial response | 158 | 157
  Stable disease | 30 | 27
  Progressive disease | 12 | 15
  Indeterminate | 15 | 22

6. Secondary Outcome: Number of Participants With Best Overall Response (BOR) Based on Investigator Assessment
Description: as for outcome 5
Time Frame: Day 28 of Cycle 1, Cycle 2 then every 8 weeks until disease progression (up to 48 months)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
Participants
  Complete response | 2 | 1
  Partial response | 169 | 157
  Stable disease | 38 | 49
  Progressive disease | 9 | 11
  Indeterminate | 9 | 7

7. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as time from first documentation of objective response(CR or PR, whichever occurred first)to date of PD/death from any cause, whichever occurred first. CR: disappearance of all target lesions (TLs), non TLs; any pathological lymph nodes (LN) must reduce in short axis to <10 mm; normalization of tumour marker level, for non TL all LN must be non-pathological in size (<10 mm short axis); PR:>=30% decrease in sum of diameters of TLs, referring baseline sum diameters. PD:>=20% increase in sum of diameters of TLs, referring smallest sum on study, sum must be an absolute increase of >=5 mm, appearance of >=1 new lesions; unequivocal progression of existing non TLs. DoR was recorded based on IRC review and investigator's assessment and summarized for subgroup of participants with objective disease response.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
months
  DoR: IRC review: number analyzed (Participants) | 170 | 161
  DoR: IRC review | 14.8 [12.0 to 17.4] | 8.3 [7.4 to 9.2]
  DoR: Investigator assessment: number analyzed (Participants) | 171 | 158
  DoR: Investigator assessment | 15.9 [13.8 to 17.6] | 9.2 [8.2 to 11.0]
Statistical Analysis 1: Comparison: Dacomitinib vs Gefitinib; Comparison of dacomitinib vs gefitinib based on IRC review; Test type: Superiority; p < 0.0001, 1-sided stratified log-rank test; Hazard Ratio (HR) = 0.403, 95% CI 2-sided [0.307 to 0.529] — Based on stratified Cox regression model
Statistical Analysis 2: Comparison: Dacomitinib vs Gefitinib; Comparison of dacomitinib vs gefitinib based on Investigator assessment; Test type: Superiority; p < 0.0001, 1-sided stratified log-rank test; Hazard Ratio (HR) = 0.545, 95% CI 2-sided [0.418 to 0.711] — Based on stratified Cox regression model

8. Secondary Outcome: Objective Response Rate (ORR) Based on IRC Review
Description: Percentage of participants with a BOR of either CR or PR based on IRC review recorded from the start of treatment until disease progression based on RECIST v1.1. CR: disappearance of all target lesions (TLs), non TLs; any pathological lymph nodes (LN) must reduce in short axis to <10 mm; normalization of tumour marker level, for non TL all LN must be non-pathological in size (<10 mm short axis); PR:>=30% decrease in sum of diameters of TLs, referring baseline sum diameters. PD:>=20% increase in sum of diameters of TLs, referring smallest sum on study, sum must be an absolute increase of >=5 mm, appearance of >=1 new lesions; unequivocal progression of existing non TLs.
Time Frame: Day 28 of Cycle 1, Cycle 2 then every 8 weeks until disease progression (up to 48 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
percentage of participants | 74.9 [68.7 to 80.4] | 71.6 [65.2 to 77.4]
Statistical Analysis 1: Comparison: Dacomitinib vs Gefitinib; Test type: Superiority; p = 0.1942, Cochran-Mantel-Haenszel

9. Secondary Outcome: Objective Response Rate (ORR) Based on Investigator Assessment
Description: Percentage of participants with a BOR of either CR or PR based on investigator assessment recorded from the start of treatment until disease progression based on RECIST v1.1. CR: disappearance of all target lesions (TLs), non TLs; any pathological lymph nodes (LN) must reduce in short axis to <10 mm; normalization of tumour marker level, for non TL all LN must be non-pathological in size (<10 mm short axis); PR:>=30% decrease in sum of diameters of TLs, referring baseline sum diameters. PD:>=20% increase in sum of diameters of TLs, referring smallest sum on study, sum must be an absolute increase of >=5 mm, appearance of >=1 new lesions; unequivocal progression of existing non TLs.
Time Frame: Day 28 of Cycle 1, Cycle 2 then every 8 weeks until disease progression (up to 48 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 225
percentage of participants | 75.3 [69.2 to 80.8] | 70.2 [63.8 to 76.1]
Statistical Analysis 1: Comparison: Dacomitinib vs Gefitinib; Test type: Superiority; p = 0.0924, Cochran-Mantel-Haenszel

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.AEs included both serious and non- serious adverse events. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs were events between first dose of study drug and up to 28-35 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From randomization until death or last date known as alive, up to 91 months
Population: Safety analysis set included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Dacomitinib (Ongoing at DCO): DCO was the protocol-defined cutoff at 48 months from first dosing of the last enrolled participant (13 May 2019). At the DCO, 11 participants were ongoing in the dacomitinib arm and continued study treatment until disease progression, intolerable toxicities, withdrawal, death, or study terminated by sponsor, whichever occurred first. The 11 participants were analyzed for adverse events after LPLV on 27 Jan 2022.
Arm/Group | Dacomitinib | Gefitinib | Dacomitinib (Ongoing at DCO)
Number analyzed (Participants) | 227 | 224 | 11
Participants
  TEAEs | 226 | 220 | 11
  SAEs | 69 | 53 | 4

11. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities of Grade 3 or Higher Severity Based on NCI CTCAE Version 4.03: Biochemistry and Haematology
Description: Parameters included anaemia, activated partial thromboplastin time, haemoglobin, international normalized ratio, lymphocyte count, lymphopenia, neutrophils (absolute), platelets, prothrombin time and white blood cells. Biochemistry parameters included alanine aminotransferase (increased), alkaline phosphatase (increased), aspartate aminotransferase (increased), bilirubin (total), creatinine (increased), hypercalcaemia, hyperglycaemia, hyperkalaemia, hypermagnesaemia, hypernatraemia, hypoalbuminaemia, hypocalcaemia, hypoglycaemia, hypokalaemia, hypomagnesaemia, hyponatraemia. Test abnormalities were graded by AEs according to the Common Terminology Criteria for Adverse Events(NCI CTCAE) version 4.03 as Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening; Grade 5=death related to AE. Only categories with at least 1 participant with abnormality are reported in this outcome measure.
Time Frame: From randomization until death or last date known as alive, up to 61 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 224
Participants
  Anaemia (Grade 3) | 5 | 6
  Haemoglobin increased(Grade 3) | 0 | 1
  Lymphopenia (Grade 3) | 13 | 6
  Neutrophil count (absolute) (Grade 3) | 0 | 2
  WBC count (Grade 3) | 1 | 1
  Alanine aminotransferase increased (Grade 3) | 5 | 26
  Alanine aminotransferase increased (Grade 4) | 0 | 3
  Aspartate aminotransferase increased (Grade 3) | 2 | 15
  Aspartate aminotransferase increased (Grade 4) | 0 | 3
  Alkaline phosphatase increased (Grade 3) | 2 | 5
  Bilirubin increased (total) (Grade 3) | 1 | 1
  Creatinine increased (Grade 3) | 1 | 1
  Hypercalcemia (Grade 3) | 1 | 0
  Hyperglycemia (Grade 3) | 2 | 5
  Hyperkalemia (Grade 3) | 0 | 1
  Hyperkalemia (Grade 4) | 0 | 2
  Hypermagnesemia (Grade 3) | 9 | 7
  Hypocalcemia (Grade 3) | 3 | 4
  Hypoglycemia (Grade 3) | 0 | 2
  Hypoglycemia (Grade 4) | 1 | 0
  Hypokalemia (Grade 3) | 13 | 5
  Hypokalemia (Grade 4) | 2 | 0
  Hypomagnesemia (Grade 3) | 2 | 0
  Hyponatremia (Grade 3) | 5 | 4
  Hyponatremia (Grade 4) | 1 | 1

12. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities: Urinalysis
Description: Urinalysis parameter included urine protein, urine blood/haemoglobin, urine glucose and urine sediment. Test abnormalities was defined as deviation from normal range (higher or lower). Normal range of 24-hour urine protein test: less than 150 mg of protein per day, urine glucose: 0 to 0.8 mmol/L (millimole per liter), urine protein: 0 to 20 mg/dL (milligrams per deciliter). Urine blood/haemoglobin abnormality was defined as presence and absence of blood/haemoglobin in urine of participants. Urine sediment abnormality was defined as the presence of any bacteria, casts, crystals, and epithelial cells. Only categories with at least 1 participant with abnormality are reported in this outcome measure.
Time Frame: From randomization until death or last date known as alive, up to 61 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 224
Participants
  High Urine Protein | 1 | 1
  Low Urine Glucose | 1 | 0
  High Urine Blood/Haemoglobin | 4 | 4

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Criteria for vital signs abnormalities: postbaseline pulse rate less than (<) 50 beats per minute (bpm) or greater than (>)130 bpm and maximum increase from baseline in pulse rate >=30 bpm and maximum decrease from baseline in pulse rate <=30 bpm. Systolic blood pressure (BP) of maximum increase from baseline (MIB) >=40 millimeters of mercury (mmHg), maximum decrease from baseline (MDB) in systolic blood pressure =<60 mmHg. Diastolic blood pressure of MIB >=20 mmHg and MDB in diastolic blood pressure >-40 and =<-20 mm Hg. And MDB in diastolic BP<=-40 mmHg. Only categories with at least 1 participant with abnormality are reported in this outcome measure.
Time Frame: From randomization until death or last date known as alive, up to 61 months
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 227 | 224
Participants
  MIB in systolic BP >=40 mmHg: number analyzed (Participants) | 224 | 223
  MIB in systolic BP >=40 mmHg | 16 | 22
  MDB in systolic BP <=-60 mmHg: number analyzed (Participants) | 224 | 223
  MDB in systolic BP <=-60 mmHg | 0 | 1
  MIB in diastolic BP >=20 mmHg: number analyzed (Participants) | 224 | 223
  MIB in diastolic BP >=20 mmHg | 42 | 44
  MDB in diastolic BP >-40 and <=-20mmHg: number analyzed (Participants) | 224 | 223
  MDB in diastolic BP >-40 and <=-20mmHg | 51 | 53
  MDB in diastolic BP <=-40 mmHg: number analyzed (Participants) | 224 | 223
  MDB in diastolic BP <=-40 mmHg | 0 | 1
  Maximum post baseline pulse rate >130 bpm: number analyzed (Participants) | 226 | 223
  Maximum post baseline pulse rate >130 bpm | 2 | 2
  Minimum post baseline pulse rate <50 bpm: number analyzed (Participants) | 226 | 223
  Minimum post baseline pulse rate <50 bpm | 3 | 0
  MIB in pulse rate >=30 bpm: number analyzed (Participants) | 225 | 223
  MIB in pulse rate >=30 bpm | 16 | 12
  MDB in pulse rate <=-30 bpm: number analyzed (Participants) | 225 | 223
  MDB in pulse rate <=-30 bpm | 17 | 15
  MIB in body weight >=10%: number analyzed (Participants) | 225 | 223
  MIB in body weight >=10% | 28 | 42
  MDB in body weight <=-10%: number analyzed (Participants) | 225 | 223
  MDB in body weight <=-10% | 46 | 32

14. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Electrocardiogram (ECG)
Description: ECG parameters included corrected QT interval using Bazett's formula (QTcB) and corrected QT interval using Fridericia's formula (QTcF). ECG criteria for abnormality: absolute value 450 - <480 msec, 480 - <500 msec, >=500msec. The number of participants with potentially clinically significant ECG findings at any visit were reported.
Time Frame: From randomization until death or last date known as alive, up to 61 months
Population: Safety analysis set included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received. Here, "N" (number of participants analyzed) signifies participants who were evaluable for this specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 217 | 7
Participants
  QTcF Criteria: 450-<480 | 5 | 0
  QTcB Criteria: 450-<480 | 22 | 0
  QTcB Criteria: 480-<500 | 3 | 0

15. Secondary Outcome: Number of Participants With Maximum Relative Decrease From Baseline >20% in Left Ventricular Ejection Fraction (LVEF)
Description: An ejection fraction (EF) was the volumetric fraction of blood ejected from a ventricle of the heart with each heartbeat; it was a measure of the pumping efficiency of the heart. The EF of the left heart, known as the left ventricular ejection fraction, was a measure of the efficiency of pumping into the body's systemic circulation.
Time Frame: From baseline up to 7 days of Cycle 4 (up to 91 days)
Population: Safety analysis set included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received. Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 191 | 199
Participants | 5 | 5

16. Secondary Outcome: Health Related Quality of Life (HRQOL): Time to Deterioration (TTD) in Pain, Dyspnea, Fatigue or Cough
Description: HRQOL was measured by standardized questionnaires (European Organization for Research and Treatment of Cancer (EORTC)) quality of life questionnaires (OLQ-C30) and its lung cancer module (QLQ-LC13). TTD in pain (chest, arm/shoulder), dyspnea, fatigue or cough was defined as time between baseline and first occurrence of increase in score of 10 points or greater from baseline in any of these 4 symptoms for at least two consecutive cycles. For those who had not shown deterioration, the data was censored at the last date when the participants completed an assessment for pain, dyspnea, fatigue or cough.
Time Frame: Baseline until the end of treatment (up to 48 months)
Population: Patient reported outcomes (PRO) analysis set included all enrolled participants, who started treatment and completed a baseline PRO assessments and at least one post-baseline PRO assessment after the first dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 226 | 222
months | 3.8 [2.3 to 4.8] | 6.6 [3.8 to 9.3]
Statistical Analysis 1: Comparison: Dacomitinib vs Gefitinib; Test type: Superiority; p = 0.1641, Unstratified Log-rank Test; Cox Proportional Hazard = 1.173, 95% CI 2-sided [0.928 to 1.483]

17. Secondary Outcome: Overall Mean Scores of Euro Quality of Life-5 Dimension Visual Analog Scale (EQ-5D VAS)
Description: The Euro Quality of Life-5 dimension (EQ-5D) is a brief self-administered, validated reliable generic health status instrument. EQ-5D general health status can also be measured by a visual analog scale (EQ-5D VAS). EQ-5D VAS measures the participant's self-rated health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: From Cycle 1 Day 1 up to 48 months
Population: PRO analysis set included all enrolled participants, who started treatment and completed a baseline PRO assessments and at least one post-baseline PRO assessment after the first dose. Here "N" signifies number of participants who were evaluable for this specified outcome measure.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dacomitinib | Gefitinib
Number analyzed (Participants) | 224 | 221
units on a scale | 73.3869 [71.608 to 75.166] | 77.6923 [75.895 to 79.490]

18. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Dacomitinib and Its Metabolite PF-05199265
Description: Cmax was defined as maximum observed plasma concentration and can be observed directly from data.
Time Frame: Pre-dose and 2, 4, 6, 8, and 24 hours post-dose on Cycle 2 Day 1 (Day 29)
Population: Pharmacokinetic (PK) analysis set included all participants who were treated with dacomitinib with at least 1 measured plasma concentration and were dose-compliant (who received 45 mg dacomitinib daily without interruptions/dose reductions for at least 14 days prior to day of data collection). This outcome measure was planned to be analyzed in Chinese subgroup only.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Dacomitinib
Number analyzed (Participants) | 19
nanogram per milliliter (ng/mL)
  Dacomitinib | 84.19 (21.90)
  PF-05199265 | 12.77 (7.58)

19. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Dacomitinib and Its Metabolite PF-05199265
Description: Tmax was defined as time to first occurrence of Cmax and can be observed directly from data as time of first occurrence.
Time Frame: Pre-dose and 2, 4, 6, 8, and 24 hours post-dose (sample collection time points had window of +/- 10% of nominal time) on Cycle 2 Day 1 (Day 29)
Population: PK analysis set included all participants who were treated with dacomitinib with at least 1 measured plasma concentration and were dose-compliant (who received 45 mg dacomitinib daily without interruptions/dose reductions for at least 14 days prior to day of data collection). This outcome measure was planned to be analyzed in Chinese subgroup only.
Measure: Median (Full Range); unit: hour
Arm/Group | Dacomitinib
Number analyzed (Participants) | 19
hour
  Dacomitinib | 4.03 [2.0 to 24.0]
  PF-05199265 | 6.0 [0.0 to 25.0]

20. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero (0) to End of Dosing Interval (AUCtau) of Dacomitinib and Its Metabolite PF-05199265
Description: AUCtau was defined as area under the plasma concentration-time curve over dosing interval tau and was determined by Linear/Log trapezoidal method.
Time Frame: Pre-dose and 2, 4, 6, 8, and 24 hours post-dose on Cycle 2 Day 1 (Day 29)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Dacomitinib
Number analyzed (Participants) | 19
nanogram*hour/milliliter (ng*hr/mL)
  Dacomitinib | 1712.08 (413.61)
  PF-05199265 | 278.47 (163.53)

21. Secondary Outcome: Averaged Plasma Concentration at Steady State (Cavg) of Dacomitinib and Its Metabolite PF-05199265
Description: Cavg was defined as averaged plasma concentration at steady state, and was calculated as AUCtau/tau.
Time Frame: Pre-dose and 2, 4, 6, 8, and 24 hours post-dose on Cycle 2 Day 1 (Day 29)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dacomitinib
Number analyzed (Participants) | 19
ng/mL
  Dacomitinib | 71.33 (17.23)
  PF-05199265 | 11.60 (6.81)

22. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of Dacomitinib and Its Metabolite PF-05199265
Description: Cmin was defined as minimum observed plasma concentration and can be observed directly from data.
Time Frame: Pre-dose and 2, 4, 6, 8, and 24 hours post-dose on Cycle 2 Day 1 (Day 29)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dacomitinib
Number analyzed (Participants) | 19
ng/mL
  Dacomitinib | 60.64 (14.85)
  PF-05199265 | 10.49 (6.26)

23. Secondary Outcome: Fluctuation Coefficient Between Trough and Peak Plasma Concentration (DF) of Dacomitinib and Its Metabolite PF-05199265
Description: Fluctuation coefficient between trough and peak plasma concentration was determined as Cmax-Ctrough divided by Cavg, where Cmax was the maximum observed concentration within the dosing interval, Ctrough was the observed concentration prior to dose administration and Cavg was averaged plasma concentration at steady state.
Time Frame: Pre-dose and 2, 4, 6, 8, and 24 hours post-dose on Cycle 2 Day 1 (Day 29)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Fluctuation coefficient
Arm/Group | Dacomitinib
Number analyzed (Participants) | 19
Fluctuation coefficient
  Dacomitinib | 0.2883 (0.1460)
  PF-05199265 | 0.1105 (0.0827)

24. Secondary Outcome: Apparent Clearance (CL) of Dacomitinib
Description: Drug clearance was a quantitative measure of the rate at which a drug substance was removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes).
Time Frame: Pre-dose and 2, 4, 6, 8, and 24 hours post-dose on Cycle 2 Day 1 (Day 29)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | Dacomitinib
Number analyzed (Participants) | 19
Liter/hour | 27.61 (5.97)

25. Secondary Outcome: Pre-dose Plasma Concentrations (Ctrough) of Dacomitinib and Its Metabolite PF-05199265
Description: Trough plasma concentration was defined as the measured concentration at the end of a dosing interval at steady state (taken directly before next administration).
Time Frame: Pre-dose on Day 1 of Cycle 2, 3, 4, 5 and 6
Population: PK analysis set included all participants who were treated with dacomitinib with at least one measured plasma concentration and were dose-compliant. Dose-compliant participants were those who received 45 mg dacomitinib daily without interruptions or dose reductions for at least 14 days prior to the day of data collection. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dacomitinib
Number analyzed (Participants) | 188
ng/mL
  Cycle 2 Day 1: Dacomitinib: number analyzed (Participants) | 176
  Cycle 2 Day 1: Dacomitinib | 70.24 (27.16)
  Cycle 3 Day 1: Dacomitinib: number analyzed (Participants) | 143
  Cycle 3 Day 1: Dacomitinib | 68.34 (25.80)
  Cycle 4 Day 1: Dacomitinib: number analyzed (Participants) | 112
  Cycle 4 Day 1: Dacomitinib | 68.16 (25.49)
  Cycle 5 Day 1: Dacomitinib: number analyzed (Participants) | 85
  Cycle 5 Day 1: Dacomitinib | 64.50 (25.52)
  Cycle 6 Day 1: Dacomitinib: number analyzed (Participants) | 74
  Cycle 6 Day 1: Dacomitinib | 61.68 (22.58)
  Cycle 2 Day 1: PF-05199265: number analyzed (Participants) | 176
  Cycle 2 Day 1: PF-05199265 | 13.20 (8.55)
  Cycle 3 Day 1: PF-05199265: number analyzed (Participants) | 143
  Cycle 3 Day 1: PF-05199265 | 14.42 (9.10)
  Cycle 4 Day 1: PF-05199265: number analyzed (Participants) | 112
  Cycle 4 Day 1: PF-05199265 | 13.70 (8.33)
  Cycle 5 Day 1: PF-05199265: number analyzed (Participants) | 85
  Cycle 5 Day 1: PF-05199265 | 12.48 (6.69)
  Cycle 6 Day 1: PF-05199265: number analyzed (Participants) | 74
  Cycle 6 Day 1: PF-05199265 | 13.05 (6.52)

ADVERSE EVENTS:
Time Frame: From randomization until death or last date known as alive, up to 91 months
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety analysis set included all participants who received at least 1 dose of study medication, with treatment assignments designated according to actual study treatment received.
Arm/Group | Dacomitinib | Gefitinib | Dacomitinib (Ongoing at DCO)
All-Cause Mortality (participants affected / at risk) | 133/227 | 152/224 | 1/11
Serious Adverse Events (participants affected / at risk) | 69/227 | 53/224 | 4/11
Other Adverse Events (participants affected / at risk) | 224/227 | 217/224 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib (N=227) | Gefitinib (N=224) | Dacomitinib (Ongoing at DCO) (N=11)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 9 | 12 | 0
Death (General disorders) | 1 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 2 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 3 | 0
Cerebral venous thrombosis (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 0 | 1
Otitis media chronic (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dacomitinib (N=227) | Gefitinib (N=224) | Dacomitinib (Ongoing at DCO) (N=11)
Anaemia (Blood and lymphatic system disorders) | 27 | 18 | 5
Diarrhoea (Gastrointestinal disorders) | 199 | 125 | 10
Stomatitis (Gastrointestinal disorders) | 99 | 41 | 6
Nausea (Gastrointestinal disorders) | 45 | 50 | 3
Constipation (Gastrointestinal disorders) | 32 | 29 | 2
Mouth ulceration (Gastrointestinal disorders) | 32 | 14 | 3
Vomiting (Gastrointestinal disorders) | 22 | 29 | 0
Aphthous ulcer (Gastrointestinal disorders) | 13 | 6 | 0
Oral pain (Gastrointestinal disorders) | 13 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 14 | 13 | 0
Dysphagia (Gastrointestinal disorders) | 10 | 12 | 1
Abdominal pain upper (Gastrointestinal disorders) | 10 | 14 | 0
Asthenia (General disorders) | 32 | 30 | 1
Chest pain (General disorders) | 19 | 27 | 3
Fatigue (General disorders) | 26 | 20 | 1
Mucosal inflammation (General disorders) | 21 | 8 | 0
Pyrexia (General disorders) | 22 | 18 | 3
Oedema peripheral (General disorders) | 13 | 7 | 0
Pain (General disorders) | 16 | 14 | 3
Paronychia (Infections and infestations) | 140 | 45 | 9
Conjunctivitis (Infections and infestations) | 46 | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 36 | 29 | 5
Nasopharyngitis (Infections and infestations) | 26 | 20 | 3
Rash pustular (Infections and infestations) | 15 | 3 | 2
Urinary tract infection (Infections and infestations) | 14 | 8 | 0
Weight decreased (Investigations) | 67 | 43 | 5
Alanine aminotransferase increased (Investigations) | 53 | 90 | 7
Aspartate aminotransferase increased (Investigations) | 49 | 84 | 5
Blood bilirubin increased (Investigations) | 19 | 20 | 1
Blood alkaline phosphatase increased (Investigations) | 16 | 8 | 2
Gamma-glutamyltransferase increased (Investigations) | 17 | 19 | 3
White blood cell count decreased (Investigations) | 6 | 14 | 1
Weight increased (Investigations) | 11 | 19 | 3
Decreased appetite (Metabolism and nutrition disorders) | 73 | 58 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 25 | 13 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 26 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 26 | 31 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 37 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 14 | 2
Dysgeusia (Nervous system disorders) | 15 | 11 | 0
Paraesthesia (Nervous system disorders) | 15 | 11 | 1
Headache (Nervous system disorders) | 17 | 21 | 1
Dizziness (Nervous system disorders) | 12 | 17 | 2
Insomnia (Psychiatric disorders) | 32 | 33 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 46 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 29 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 5 | 3
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 15 | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 10 | 13 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 12 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 112 | 64 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 64 | 39 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 53 | 29 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 47 | 33 | 3
Rash (Skin and subcutaneous tissue disorders) | 41 | 26 | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 33 | 7 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 29 | 27 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 25 | 9 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 21 | 7 | 1
Acne (Skin and subcutaneous tissue disorders) | 19 | 13 | 0
Erythema (Skin and subcutaneous tissue disorders) | 14 | 3 | 1
Hypertension (Vascular disorders) | 19 | 21 | 2
Dry eye (Eye disorders) | 12 | 8 | 3
Angular cheilitis (Gastrointestinal disorders) | 12 | 2 | 0
Folliculitis (Infections and infestations) | 12 | 4 | 1
Haemoglobin decreased (Investigations) | 14 | 5 | 0
Blood lactate dehydrogenase increased (Investigations) | 8 | 12 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 10 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 8 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 2
Corneal erosion (Eye disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Trichiasis (Eye disorders) | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1
Mass (General disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Immune system disorder (Immune system disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 2
Nasal vestibulitis (Infections and infestations) | 0 | 0 | 2
Gingivitis (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 3
Blood albumin decreased (Investigations) | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 0 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Tetany (Metabolism and nutrition disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1
Vertebral artery stenosis (Nervous system disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 0 | 1
Vulvovaginal rash (Reproductive system and breast disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ischaemia (Vascular disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.